CLINICAL TRIAL: NCT07359885
Title: Prediction of Postoperative Pulmonary Complications in Thoracic Surgery: an Immuno-inflammatory Approach
Brief Title: Prediction of Postoperative Pulmonary Complications in Thoracic Surgery
Acronym: PREDICT-PPC
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2024/0307/HP; 2025-A01699-40 (Other: ANSM)
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Pulmonary Complications (PPCs)
Keywords: lung cancer; immuno-inflammatory approach
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — Additional samples, taken as part of routine care, of 2 x 5 mL of blood in heparinized tubes taken at visits V1, V2 and V3
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Evaluation of prognostic performance of a defined score using a machine learning method (STABL: Stability Selection) integrating immune data (cytometric and proteomic) — Determination of the area under the curve (AUC) Receiver Operating Curve (ROC) for predicting complications calculated from the score obtained by the machine learning method and the occurrence of at least one major pulmonary complication among the following in the first 7 postoperative days: postoperative pneumonia, pleural effusion, postoperative atelectasis, pneumothorax, bronchospasm and acute respiratory distress syndrome.

SUMMARY:
Lung cancer is a common disease, and its treatment is lobectomy or pulmonary segmentectomy. In France, approximately 8,000 patients undergo this procedure each year, but it remains associated with significant Postoperative Pulmonary Complications (PPC). This surgical trauma triggers a multicellular and orchestrated immune response, necessary for defense against pathogens, as well as for inflammatory resolution and wound healing. Preoperative single-cell analysis of the patient's immune system is therefore a promising strategy for identifying biomarkers of postoperative pulmonary complications (PPC). Brice Gaudilliere's laboratory at Stanford University, in collaboration with the Paris-based startup Surge, has developed and patented a multivariate model integrating mass cytometry data, proteomic analyses, and clinical data collected before surgery to accurately predict surgical site complications after major abdominal surgery. However, no study has yet explored the identification of inflammatory biomarkers predictive of PPC after thoracic surgery.

DETAILED DESCRIPTION:
The issue of postoperative pulmonary complications following major lung resection (such as lobectomy or segmentectomy) is a central topic in anesthesia and thoracic surgery. Postoperative morbidity and mortality after this type of surgery have drastically decreased in recent years with advances in anesthesia and resuscitation, as well as minimally invasive surgery, but remain high compared to other types of surgery, particularly due to postoperative pneumonia. The etiology of postoperative pneumonia is multifactorial (atelectasis, postoperative ventilation, inadequate analgesia), but the patient's immune system plays a predominant role in each individual case. Therefore, identifying inflammatory biomarkers predictive of postoperative pulmonary complications in a given patient could optimize their management and reduce the risk of postoperative pulmonary cancer (PPC). The objective of this study is to identify preoperative inflammatory biomarkers predictive of PPC after major lung resection. It will use machine learning methods specific to these data to define an immune signature of PPC. This immune signature will be validated using standard analytical techniques to facilitate the clinical translation of a diagnostic test.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* ASA score ≤ 3
* Patients undergoing scheduled video-assisted or robot-assisted lobectomy, bilobectomy, or segmentectomy.
* Patients who have read and understood the information letter and do not object to the research.
* For women of childbearing age (non-sterile): effective contraception
* Menopausal (non-medically induced amenorrhea for at least 12 months)
* Patients covered by a social security scheme

Exclusion Criteria:

* Minor patients
* Surgery scheduled for a Friday
* Patients undergoing a pneumonectomy
* Pregnant or breastfeeding women
* Patients deprived of their liberty by an administrative or judicial decision, as well as those under legal protection, guardianship, or curatorship

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing programmed video-assisted or robot-assisted lobectomy, bilobectomy or segmentectomy.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the prognostic performance of a score for screening patients at risk of postoperative pulmonary complications (PPC) | Evaluation of the prognostic performance of a defined score using a machine learning method (STABL: Stability Selection) integrating preoperative immune (cytometric and proteomic) and clinical data within 7 postoperative days of a major lung resection

SECONDARY OUTCOMES:
Evaluation of the incidence of pulmonary complications | 30 days
  Postoperative Pulmonary Complications (PPCs) occurring between the 8th and 30th postoperative days will be assessed. The PPCs considered will be: postoperative pneumonia, pleural effusion, postoperative atelectasis, pneumothorax, bronchospasm, and acute respiratory distress syndrome.
Evaluation of the correlation between the prognostic score defined using a machine learning method and the length of hospital stay | 3 months
  Measurement of the score obtained by the machine learning method and the length of hospital stay recorded in days (D0 being the day of the intervention)
Evaluation of the correlation between the prognostic score defined using a machine learning method and the number of reintubations recorded | 30 days
  Measurement of the score obtained by the machine learning method and the number of reintubations recorded in the first 30 postoperative days
Evaluation of the correlation between the prognostic score defined using a machine learning method and the Number of unplanned hospitalizations in intensive care recorded | 30 days
  Measurement of the score obtained by the machine learning method and the Number of unplanned hospitalizations in intensive care recorded in the first 30 postoperative days
Evaluation of the correlation between the prognostic score defined using a machine learning method and the Preoperative anxiety score assessed | 48 hours
  Measurement of the score obtained by the machine learning method and the Preoperative anxiety score assessed on day 0 (before surgery) using the STAI (State Trait Anxiety Inventory) Questionnaire
Evaluation of the correlation between the prognostic score defined using a machine learning method and the Preoperative anxiety score assessed | 48 hours
  Measurement of the score obtained by the machine learning method and the Preoperative anxiety score assessed at 48 hours using the STAI (State Trait Anxiety Inventory) Questionnaire
Evaluation of the correlation between the prognostic score defined using a machine learning method and The cost of care | 3 months
  Measurement of the score obtained by the machine learning method and The cost of care between J0, J30 and J90 (estimated by the Homogeneous Stay Group generated for each hospital stay (initial hospitalization and rehospitalization(s)).
Evaluation of the prognostic performance of the score calculated by the machine learning method on Post-operative Pulmonary Complications (PPC) assessed by the Melbourne composite score (Melbourne Group Scale (MGS) >=4) | 7 days
  The area under the receiver operating curve (AUC) is calculated from the score obtained using the machine learning method and the primary respiratory symptoms (PRS) in the first 7 days, assessed by the Melbourne Group Scale (MGS).
  The MGS includes the following items and will be considered positive if ≥ 4 points:
  Temperature ≥ 38.5°C (1 point) Purulent sputum (1 point) Positive bacteriology (1 point) SpO2 < 90% in room air (1 point) Leukocytes > 11.2 x 10⁶/ml (1 point) Prescription of antibiotic therapy (1 point) Chest X-ray: atelectasis (1 point) (defined as previously) Diagnosis of pneumonia by a physician (1 point) (defined as previously) Readmission to intensive care or prolonged stay (> 36 hours) for respiratory problems (1 point)
Evaluation of the prognostic performance of the score calculated by the machine learning method on the severity of postpartum bleeding (PPB) | 30 days
  The area under the receiver operating curve (AUC) is calculated from the score obtained using the machine learning method and the severity of postpartum bleeding (PPB) in the first 30 days assessed by the Clavien-Dindo score
Evaluation of the prognostic performance of the score calculated by the machine learning method on Postoperative mortality assessed at 30 days | 30 days
  The area under the receiver operating curve (AUC) is calculated from the score obtained using the machine learning method and Postoperative mortality assessed at 30 days
Evaluation of the prognostic performance of the score calculated by the machine learning method on Postoperative mortality assessed at 90 days | 90 days
  The area under the receiver operating curve (AUC) is calculated from the score obtained using the machine learning method and Postoperative mortality assessed at 90 days
Evaluation of the prognostic performance of the score calculated by the machine learning method on Pre- and postoperative pain | 90 days
  The area under the receiver operating curve (AUC) is calculated from the score obtained using the machine learning method and Pre- and postoperative pain was assessed using a numerical rating scale from 0 to 10 at day 0 (before surgery), at 24 hours, and at 48 hours. Neuropathic pain was assessed by telephone at 3 months using the DN4 questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Jean JS SELIM, Doctor, Study Director — Service de Anesthésie-Réanimation Médecine périopératoire CHU de Rouen
Locations (1):
- Service de Anesthésie-Réanimation Médecine périopératoire CHU de Rouen, Rouen, France

IPD SHARING:
Plan to Share IPD: No